CLINICAL TRIAL: NCT04066556
Title: Prospective Multicenter Registry for Acute Ischemic Stroke Patients With Standard Reperfusion Therapy
Brief Title: SMART-EST(Specialized Multi-center Attributed Registry of sTroke - EndovaScular or Thrombolytic Therapy)
Status: Active, not recruiting | Type: Observational
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Other Study IDs: 4-2019-0486
Record Dates: First submitted 2019-08-21; First posted 2019-08-26 (Actual); Last update posted 2019-08-28 (Actual); Status verified 2019-08

CONDITIONS: Ischemic Stroke
Keywords: Stroke; Recanalization treatment; Outcome; Collateral; Thrombus; CT; Comorbidity
MeSH Terms: conditions — Ischemic Stroke; Stroke; Thrombosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 10 Years
Biospecimen Retention: Samples With DNA — whole blood, frozen tissue
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Acute ischemic stroke patients: Acute ischemic stroke patients who received intravenous (IV) thrombolysis and/or intra-arterial (IA) recanalization treatment
  Interventions: Other: Brain CT imaging

INTERVENTIONS:
Other: Brain CT imaging — The investigators will analyzed the CT image that was performed in patients with hyperacute stroke. The CT protocol includes CT thrombus, collateral, core images. The investigators also obtain detailed history and laboratory and imaging result for comorbidity. The comorbidity index protocol is based on the Charlson comorbidity index.
  * Cut-off values in thrombus volume and Hounsfield unit according to non-contrast CT images
  * Cut-off values in areas of irreversible changes according to non-contrast CT images
  * Cut-off values in occlusion sites and collateral scores according to CT angiographies
  * Cut-off values of consolidated CT imaging index including clot, core, and collateral score
  * Cut-off values of comorbidity index
  * Medical care expenses according to comorbidity index in patients who received intravenous thrombolytic treatment and/or endovascular recanalization treatments.

SUMMARY:
Use of intravenous(IV) thrombolysis and intra-arterial(IA) recanalization treatment has been rapidly increasing, However, despite of the treatment, recanalization rates are 22.6 - 70% and only 30-50% of patients show meaningful clinical improvements. Mechanisms of futile recanalization may include 1) large ischemic core, 2) poor collateral, and 3) presence of comorbidity. In this regards, developing selection criteria using acute stroke imaging and comorbidity is warranted.

The investigators will recruit the consecutive acute stroke patients who received IV thrombolysis and/or IA recanalization treatment. This study will perform with prospective design to develop CT-based clot, core and collateral scores and a comorbidity index for selecting stroke patients who are at high risks by the treatment. The investigators will firstly establish the CT-based scores and comorbidity index using a pre-existing cohort database. Using these CT-based and comorbidity index, the investigators will validate them in a multi-center prospectively cohort.

DETAILED DESCRIPTION:
1)Full design

1. The study proceeds with a parallel design of retrospective and prospective research.
2. As in the retrospective study, this study aims to establish the ideal screening criteria and to verify the efficacy of the thrombolytic procedure by using the relevant image information, clinical information, and the history of the subjects.
3. This study is an observational study, and there is no intervention for the study.

2) retrospective design

1. Retrospective study was conducted as a multi-center retrospective cohort and intravenous thrombolysis and intraarterial thrombus according to the guidelines for stroke among patients who were admitted to neurology with stroke from January 1, 2012 to December 31, 2015 of participating hospitals. Patients who underwent surgical removal.
2. The retrospective study was performed after 3 months F / U and 6 months after confirming the medical history and clinical information taken before the thrombolysis and the accompanying disease history. Check whether or not.
3. We will establish the most ideal screening criteria and verify the efficacy of predicting the prognosis after thrombolysis using the relevant imaging information, clinical information and the accompanying disease history.
4. All data are collected using e-CRF, and CT angiography images of subjects are anonymized and sent to the host institution. The lead institution quantifies the clinical information, including CT angiographic indicators and accompanying diseases, in the dark.
5. Interim analysis will be conducted once when the retrospective study is completed.

3) prospective design

1. A prospective study is a multicenter prospective observational study, in which intravenous thrombolysis and arteries were already followed in accordance with guidelines for stroke among patients who were admitted to neurology after a stroke on November 1, 2016 (based on hospitalization date). Patients who have undergone internal thrombectomy
2. Obtain a written consent form from a study subject who meets the selection / exclusion criteria (see How to Obtain a Study Participation Consent Form), and collect the medical data including the accompanying diseases of the study subject and images taken before thrombosis (removal) treatment. do.
3. In the same way as retrospective study, confirm and confirm the image and clinical information and the accompanying disease history of the study subjects and confirm the survival after 3 months F / U and 6 months.
4. The observation period in the study is expected to take about 6 months (intravenous thrombolytic therapy and intraarterial reopening therapy, mRS indicator at 3 months after discharge and stroke, and survival at 6 months after stroke).
5. All data are collected using eCRF, and CT angiography images of subjects are anonymized and sent to the host institution. The lead institution quantifies CT angiography and associated disease indicators with blinded clinical information.
6. Screening (time of hospitalization due to stroke) Patients who had cerebrovascular pretreatment prior to intravenous thrombolysis and were able to identify comorbidities.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥20 years old
2. Acute ischemic stroke patients who underwent CT angiographies before IV thrombolysis and/or IA recanalization treatment
3. Patients who give an informed consents for participation in the study or the legal representative or immediate family give informed consent on behalf of patients in case of difficulty to decide study enrollment.

Exclusion Criteria:

1. Age <20 years old
2. Acute ischemic stroke patients who did not receive IV thrombolysis and/or IA recanalization treatment
3. No informed consents from patients

Ages: 20 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Acute ischemic stroke patients who received intravenous (IV) thrombolysis and/or intra-arterial (IA) recanalization treatment
Sampling Method: Probability Sample
Enrollment: 5000 (Estimated)
Dates: Start 2019-07-12 (Actual); Primary Completion 2029-06 (Estimated); Study Completion 2029-06 (Estimated)

PRIMARY OUTCOMES:
Modified Rankin scale scores | at 3 months
  Functional improvement after stroke at 3 months Scale range: 0(Best)~6(Worst) , Functional outcome measure in stroke. Levels of disability
  0: No symptoms at all
  1. No significant disability : despite symptoms : able to carry out all usual duties and activities.
  2. Slight disability : unable to carry out all previous activities but able to look after own affairs without assistance.
  3. Moderate disability : requiring some help, but able to walk without assistance.
  4. Moderate severe disability : unable to walk without assistance, and unable to attend to own bodily needs without assistance.
  5. Severe disability : bedridden, incontinent and requiring constant nursing care and attention.
  6. Death
Any death | within 6 months
  Any death within 6 months
National Institutes of Health Stroke Scale (NIHSS) scores | at 1 day
  Primary Outcome Description: Neurological improvement according to NIHSS scores National Institutes of Health Stroke Scale (NIHSS) scores
  The National Institutes of Health Stroke Scale, or NIH Stroke Scale (NIHSS) is a tool used by healthcare providers to objectively quantify the impairment caused by a stroke. The NIHSS is composed of 11 items, each of which scores a specific ability between a 0 and 4. For each item, a score of 0 typically indicates normal function in that specific ability, while a higher score is indicative of some level of impairment.The individual scores from each item are summed in order to calculate a patient's total NIHSS score. The maximum possible score is 42, with the minimum score being a 0. (total score : 0(good)~ 42(death))
Recanalization rate | at 24 hours ± 8 hours
  Recanalization rate after thrombolytic treatments in MRA, CTA, or digital subtraction angiography (DSA) at 24 hours ± 8 hours
Asymptomatic hemorrhagic transformation rate | at 24 hours ± 8 hours
  Hemorrhagic transformation rate after thrombolysis in MR or CT at 24 hours ± 8 hours
Any complication rate including extracranial life-threatening bleeding, herniation, infection rate | within 7 days
  Any complication rate including extracranial life-threatening bleeding, herniation, infection rate within 7 days

SECONDARY OUTCOMES:
Causes of deaths | within 6 month
  Causes of deaths after thrombolytic treatments within 6 month
Stroke subtypes | within 7 days
  The Trial of ORG 10172 in Acute Stroke Treatment (TOAST) classification

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Neurology, Yonsei University College of Medicine, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: Undecided